CLINICAL TRIAL: NCT06099171
Title: Effectiveness of a Combined Therapy With Paravertebral Oxygen-ozone Injections and Topical Patch Containing Cannabidiol and β-Caryophyllene for Treatment of Neck Pain: a Prospective, Randomized, Controlled Trial.
Brief Title: Therapy With Paravertebral Oxygen-ozone Injections and Topical Cannabidiol and β-Caryophyllene Patch in Neck Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Cristiano Sconza, Principal Investigator, Humanitas Clinical and Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OZLEVOTENS
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen-Ozone Therapy plus Cannabidiol and ß-Caryophyllene Patch (Experimental): The patients will undergo 8 session of oxygen-ozone therapy, 2 per week. In each session 10 cc of a gaseous mixture of oxygen-ozone (at a concentration of 10 μg of ozone per ml of oxygen) will be injected with 6 paravertebral injections.
  For the fisrt 2 weeks of oxygen-ozone therapy patients will be asked to apply patches with local action based on Cannabidiol and ß-Caryophyllene for 8-24 hours/day for 5 days/week.
  Interventions: Drug: Cannabidiol and β-Caryophyllene Patch; Device: Oxygen-Ozone Therapy
- Oxygen-Ozone Therapy (Active Comparator): The patients will undergo 8 session of oxygen-ozone therapy, 2 per week. In each session 10 cc of a gaseous mixture of oxygen-ozone (at a concentration of 10 μg of ozone per ml of oxygen) will be injected with 6 paravertebral injections.
  Interventions: Device: Oxygen-Ozone Therapy

INTERVENTIONS:
Drug: Cannabidiol and β-Caryophyllene Patch — Cannabidiol with its decongestant activity has a soothing action in the area of application, thanks to the association with B-caryophyllene which assists its activity
  Other Names: Levotens Patch
  Arms: Oxygen-Ozone Therapy plus Cannabidiol and ß-Caryophyllene Patch
Device: Oxygen-Ozone Therapy — Ozone (O3) is a molecule consisting of 3 atoms of oxygen in a dynamically unstable structure. O3 has the capacity to modulate inflammation. O3 when in contact with human fluids and tissues rapidly reacts, generating many reactive oxygen species, as hydrogen peroxide (H2O2), superoxide ion, and hydroxyl radical (OH-). It is suggested that through moderate oxidative stress generated by these reactive byproducts, O2O3 might produce positive effects in several pathologies, including musculoskeletal affections. Moreover, O2/O3 may directly regulate prostaglandins (PGS) and bradykinin, and suppress several proinflammatory mediators, such as IL-6, IL-8 and TNF-α

SUMMARY:
The aim of this study is to compare the effectiveness of combined treatment with paravertebral oxygen-ozone injections and topical patches containing Cannabidiol and β-Caryophyllene in patients with neck pain by evaluating the following aspects:

* Reduction of pain
* Reduction of disability associated with neck pain

DETAILED DESCRIPTION:
Neck pain is a significant public health burden worldwide, with a prevalence of 2,696.5 per 100,000, and a major cause of disability, responsible for 2.56% of all years lived with disability. Many potential therapeutic interventions are available for the treatment of neck pain, including conservative therapies, minimally invasive procedures and open surgery. In particular, oxygen-ozone percutaneous injections have been tested and have proven to be well tolerated with good clinical results.

Patch cutaneous formulated with cannabidiol and β-carophyllene (Levotens®) has proven to have muscle relaxant and anti-inflammatory effects in an animal models: The tests used allow to evaluate motor performance with reference to motor coordination skills (pole test), exploration (open field test) and resistance to continuous and accelerated movement (rotarod test). These motor skills are impaired in a pain associated inflammatory response condition such as that induced by LPS (lipopolysaccharide). The CBD and BCP-based Levotens® patch placed in the area where the inflammatory stimulus is administered allows the recovery of motor function in the three types of behaviors studied.

Previous data available demonstrate a muscle relaxant action of CBD applied topically through a patch in patients suffering from TMD.

This is a randomized, controlled, prospective evaluation comparing combined treatment with paravertebral oxygen-ozone injections and topical patches containing Cannabidiol and β-Caryophyllene with only OOT. The maximum study duration for each subject will be 6 months. A total of 52 patients will be enrolled. These patients will meet specific inclusion and exclusion criteria but can be generally characterized as patients with neck pain who have been unable to achieve satisfactory pain relief with previous conservative treatments The primary study objective is to determine whether combining Levotens® Patch with OOT could lead to better early pain control than OOT alone.

1. The primary study endpoint is to establish the improvement in NRS Pain at 14 days from the start of treatment.
2. Secondary objectives of this study are:

   * Improvement in NRS pain at 1, 2, 4, 12, 36 weeks,
   * Improvement in NDI at 1, 2, 4, 12, 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain resulting from spinal pathology present for at least 1 month with or without brachial irradiation
* Cervical radiographic and/or MRI examination certifying the pathology of the spine
* Failure of previous conservative treatment (pharmacological or physiotherapy)
* Adults
* Signing of informed consent

Exclusion Criteria:

* Specific causes of neck pain (trauma, spinal deformity, fracture, neoplasia)
* Central or peripheral neurological signs
* Rheumatic diseases: diagnosis of rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis or arthritis secondary to other inflammatory diseases, chondrocalcinosis, Paget's disease or villonodular synovitis
* Neuromuscular disorders
* Presence of cognitive-behavioral deficit or psychiatric illness which, in the opinion of the investigator, could compromise patient safety or interfere with the evaluation of the effects of the treatment
* Surgery in the previous 6 months
* Cervical infiltrative treatments in the previous 4 months
* Use of orally administered systemic steroids within 2 weeks prior to screening
* Pregnant or breastfeeding women or women planning to become pregnant during the study participation period
* Known alcohol or drug dependence currently or within the past year

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 14 days
  Measure for reporting neck pain disability. It is a 10-items questionnaire; each question is scored on a 6-point scale ranging from 0 (no disability) to 5 (full disability), and these are added together to make a total score ranging from 0 to 50, which is interpreted as follows: 0 to 4= no disability, 5 to 14= mild disability, 15 to 24= moderate disability, 25 to 34= severe disability, and greater than 34 = complete disability. Evaluators can choose to provide a percentage score as a means of dealing with unanswered questions.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 1 week
  Measure of pain intensity. The scale goes from 0 (no pain) to 10 (worst pain imaginable)
Numeric Pain Rating Scale | 2 weeks
  Measure of pain intensity. The scale goes from 0 (no pain) to 10 (worst pain imaginable)
Numeric Pain Rating Scale | 4 weeks
  Measure of pain intensity. The scale goes from 0 (no pain) to 10 (worst pain imaginable)
Numeric Pain Rating Scale | 12 weeks
  Measure of pain intensity. The scale goes from 0 (no pain) to 10 (worst pain imaginable)
Numeric Pain Rating Scale | 36 weeks
  Measure of pain intensity. The scale goes from 0 (no pain) to 10 (worst pain imaginable)
Neck Disability Index | 1 week
  Measure for reporting neck pain disability. It is a 10-items questionnaire; each question is scored on a 6-point scale ranging from 0 (no disability) to 5 (full disability), and these are added together to make a total score ranging from 0 to 50, which is interpreted as follows: 0 to 4= no disability, 5 to 14= mild disability, 15 to 24= moderate disability, 25 to 34= severe disability, and greater than 34 = complete disability. Evaluators can choose to provide a percentage score as a means of dealing with unanswered questions.
Neck Disability Index | 4 weeks
  Measure for reporting neck pain disability. It is a 10-items questionnaire; each question is scored on a 6-point scale ranging from 0 (no disability) to 5 (full disability), and these are added together to make a total score ranging from 0 to 50, which is interpreted as follows: 0 to 4= no disability, 5 to 14= mild disability, 15 to 24= moderate disability, 25 to 34= severe disability, and greater than 34 = complete disability. Evaluators can choose to provide a percentage score as a means of dealing with unanswered questions.
Neck Disability Index | 12 weeks
  Measure for reporting neck pain disability. It is a 10-items questionnaire; each question is scored on a 6-point scale ranging from 0 (no disability) to 5 (full disability), and these are added together to make a total score ranging from 0 to 50, which is interpreted as follows: 0 to 4= no disability, 5 to 14= mild disability, 15 to 24= moderate disability, 25 to 34= severe disability, and greater than 34 = complete disability. Evaluators can choose to provide a percentage score as a means of dealing with unanswered questions.
Neck Disability Index | 36 weeks
  Measure for reporting neck pain disability. It is a 10-items questionnaire; each question is scored on a 6-point scale ranging from 0 (no disability) to 5 (full disability), and these are added together to make a total score ranging from 0 to 50, which is interpreted as follows: 0 to 4= no disability, 5 to 14= mild disability, 15 to 24= moderate disability, 25 to 34= severe disability, and greater than 34 = complete disability. Evaluators can choose to provide a percentage score as a means of dealing with unanswered questions.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Sconza, MD, Principal Investigator — Humanitas Clinical and Research Center
Locations (1):
- Humanitas Clinical and Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No